CLINICAL TRIAL: NCT02576704
Title: Prognostic Value of Myocardial Perfusion Heterogeneity in Normal Dual Isotope High Speed Myocardial Perfusion Imaging With a Semi Conductor Gamma Camera.
Brief Title: Prognostic Value of Myocardial Perfusion Heterogeneity in Normal SPECT Studies
Acronym: PROMETHE
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, Barone-Rochette Gilles, Professor, University Hospital, Grenoble
Other Study IDs: 2015-30
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Disease; Coronary Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: semi conductor gamma camera — we use a new mathematic technique from entropy analysis to provide precise, objective, automated quantification of perfusion heterogeneity at stress with camera SPECT. This method may be a non-invasive imaging to assess coronary microvascular dysfunction.

SUMMARY:
Myocardial perfusion imaging is an efficient tool to assess the risk of major cardiac events for patients with known or suspected coronary artery disease. If the test is normal, or if the abnormalities of perfusion represent less than 10% of the left ventricle myocardium, the patient is considered at low risk and should be managed with optimal medical treatment only.

Recently, new gamma cameras using semi-conductor detectors have been developed. Their diagnostic performances have been demonstrated and confronted with various anatomical and functional reference techniques, such as coronary angiography and FFR. The prognostic value of a normal SPECT MPI has not been specifically assessed yet.

Coronary microvascular dysfunction (CMVD) has been demonstrated to be an early marker of coronary artery disease (CAD). Preliminary data suggest that myocardial perfusion heterogeneity (a potential surrogate marker of endothelial dysfunction) can be assessed on conventional MP-SPECT, but its additive and independent prognostic value over the presence of myocardial ischemia remain unknown.

Accordingly, the purpose of this study is :

* To assess the prognostic value of a normal myocardial perfusion stress imaging using a semiconductor gamma camera with a dual isotope high speed protocol,
* To evaluate the prognostic value of myocardial perfusion heterogeneity assessed by a new automatized image processing method, in normal SPECT MPIs.

The main hypothesis is that the presence of myocardial perfusion heterogeneity is predictive of cardiovascular events in patients referred to the Nuclear Cardiology Department for routine evaluation of known or suspected CAD.

DETAILED DESCRIPTION:
SPECT imaging protocol and analysis Stress tests and SPECTs are performed according to the routine protocols in use in our center. Briefly, at peak stress, patients were injected with thallium-201. Five to 10 minutes after stress, a 5-minutes supine acquisition was performed followed by a 5-minutes prone acquisition. Subsequently, technetium-99m-sestamibi was injected, and 2 minutes later a single 5-minutes rest acquisition was performed. During stress acquisition, patients were imaged in supine and prone positions with their arms positioned over their head. The rest acquisition was only acquired in supine position. The gated SPECT studies were performed at each acquisition. Injected activity (IA) was adjusted for patient weight. For weights of <80 kg/ 80-100 kg/>100 kg, thallium-201 IAs were 74/92/111 MBq and technetium-99m-sestamibi IAs were 300/370/450 MBq, respectively. A uniform imaging pre-treatment for the reconstruction of raw myocardial perfusion imaging data was applied, and images were reconstructed and reoriented to obtain transaxial sections of the left ventricle according to the three standard cardiac planes.

In this study, we use a new mathematic technique from entropy analysis to provide precise, objective, automated quantification of perfusion heterogeneity at stress with camera SPECT. This method may be a non-invasive imaging to assess coronary microvascular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical indication for myocardial perfusion imaging

Exclusion Criteria:

* Pregnancy
* Breastfeeding women
* Myocardial perfusion abnormalities with SSS > 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study cohort Patient referred to the Nuclear Cardiology Laboratory of the University Hospital of Grenoble for myocardial perfusion imaging for diagnosis or prognosis evaluation of suspected or know coronary artery disease, whose myocardial stress imaging was normal or with Summed stress score (SSS) < or = 4.
Sampling Method: Non-Probability Sample
Enrollment: 1119 (Actual)
Dates: Start 2011-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Composite primary outcome | 3 years
  number of cardiac death or nonfatal Myocardial Infarction

SECONDARY OUTCOMES:
first composite secondary outcome | 3 years
  number of cardiac death or nonfatal Myocardial Infarction or stroke
secondary composite secondary outcome | 3 years
  number of cardiac death or nonfatal Myocardial Infarction or stroke or number of participants with myocardial revascularization
third composite secondary outcome | 3 years
  number of all death or nonfatal Myocardial Infarction
fourth composite secondary outcome | 3 years
  number of all death or nonfatal Myocardial Infarction or stroke
fifth composite secondary outcome | 3 years
  number of all death or nonfatal Myocardial Infarction or stroke or number of participants with myocardial revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Grenoble, Grenoble, Isere, France

REFERENCES:
- [Background] Verma S, Buchanan MR, Anderson TJ. Endothelial function testing as a biomarker of vascular disease. Circulation. 2003 Oct 28;108(17):2054-9. doi: 10.1161/01.CIR.0000089191.72957.ED. No abstract available. PMID 14581384
- [Background] Schindler TH, Nitzsche EU, Schelbert HR, Olschewski M, Sayre J, Mix M, Brink I, Zhang XL, Kreissl M, Magosaki N, Just H, Solzbach U. Positron emission tomography-measured abnormal responses of myocardial blood flow to sympathetic stimulation are associated with the risk of developing cardiovascular events. J Am Coll Cardiol. 2005 May 3;45(9):1505-12. doi: 10.1016/j.jacc.2005.01.040. PMID 15862426
- [Background] Johnson NP, Gould KL. Clinical evaluation of a new concept: resting myocardial perfusion heterogeneity quantified by markovian analysis of PET identifies coronary microvascular dysfunction and early atherosclerosis in 1,034 subjects. J Nucl Med. 2005 Sep;46(9):1427-37. PMID 16157524
- [Background] Hachamovitch R, Hayes SW, Friedman JD, Cohen I, Berman DS. Comparison of the short-term survival benefit associated with revascularization compared with medical therapy in patients with no prior coronary artery disease undergoing stress myocardial perfusion single photon emission computed tomography. Circulation. 2003 Jun 17;107(23):2900-7. doi: 10.1161/01.CIR.0000072790.23090.41. Epub 2003 May 27. PMID 12771008
- [Background] Barone-Rochette G, Leclere M, Calizzano A, Vautrin E, Celine GC, Broisat A, Ghezzi C, Baguet JP, Machecourt J, Vanzetto G, Fagret D. Stress thallium-201/rest technetium-99m sequential dual-isotope high-speed myocardial perfusion imaging validation versus invasive coronary angiography. J Nucl Cardiol. 2015 Jun;22(3):513-22. doi: 10.1007/s12350-014-0016-0. Epub 2014 Nov 8. PMID 25381092